CLINICAL TRIAL: NCT04580498
Title: An Open-label, Multicenter Phase II Clinical Trial of SHR-1701 With or Without Chemotherapy in the Treatment of Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: A Trial of SHR-1701 With or Without Chemotherapy in Patients With Stage III NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-205
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR-1701+Paclitaxel+carboplatin
  Interventions: Drug: SHR-1701+Paclitaxel+carboplatin
- Treatment group B (Experimental): SHR-1701
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701+Paclitaxel+carboplatin — Drug: SHR-1701 30mg/kg Drug: Paclitaxel 175mg/m2 Drug: Carboplatin AUC 5
  Arms: Treatment group A
Drug: SHR-1701 — Drug: SHR-1701 30mg/kg
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1701 with or without chemotherapy in the treatment of unresectable stage III non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent form;
* 18 to 70 years old, both male and female;
* ECOG score: 0-1
* histopathologically or cytologically confirmed, inoperable stage III squamous cell or non-squamous cell lung cancer;
* subjects who can provide fresh or archival tumor tissue;
* Measurable lesions available;
* Major organ function is basically normal;
* Non-surgically sterile female subjects of childbearing age must have a negative serum HCG test before randomization;

Exclusion Criteria:

* histologically or cytologically confirmed mixed SCLC and NSCLC;
* subjects who have malignant pleural effusion;
* Previous systemic anti-tumor therapy for NSCLC;
* Previous thoracic radiotherapy;
* Subjects who participated in other clinical trials within 4 weeks or 5 drug half-lives(whichever is shorter) before the first dose.
* Systemic immunostimulant therapy before the first dose;
* Systemic immunosuppressive therapy before the first dose or were expected to require systemic immunosuppressive drugs during the study treatment;
* Subjects with autoimmune diseases;
* Other malignant tumors other than non-small cell lung cancer within 5 years before screening;
* Known or suspected interstitial pneumonia;
* Other moderate to severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity and seriously affect respiratory function;
* Severe cardiovascular and cerebrovascular diseases;
* Clinically significant bleeding symptoms or significant bleeding tendency within 1 month before the first dose;
* Arteriovenous thrombotic events within 3 months before the first dose;
* Positive HIV test;
* Active hepatitis B or C;
* Evidence of active tuberculosis infection within 1 year before the first dose;
* Serious infection within 4 years before the first dose;
* History of attenuated live vaccination 28 days before the first dose or expected to receive attenuated live vaccination during the study;
* Major surgeries other than diagnosis or biopsy within 28 days prior to first dose;
* Previous or planned allogeneic bone marrow transplantation or solid organ transplantation;
* History of severe allergic reactions to other monoclonal antibodies/fusion proteins;
* Allergic to any component of the randomized treatment regimen;
* Female subjects who are pregnant, lactating, or planning to get pregnant during the study period;
* Subjects who has a known history of psychotropic drug abuse, alcoholism, or drug abuse
* Presence of other conditions that, in the opinion of the investigator, would make participation in this clinical trial inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From the initiation of the first dose to 3 years
  Objective response rate
EFS | From the initiation of the first dose to 3 years
  event free survival

SECONDARY OUTCOMES:
OS | From the initiation of the first dose to 3 years
  overall survival
EFS rate | From the initiation of the first dose to 3 years
  event free survival rate
TDDM | From the initiation of the first dose to 3 years
  time to death or distant metastasis
Adverse events(AEs) | From the initiation of the first dose to 90 days after the last dose
  Incidence of treatment-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China